CLINICAL TRIAL: NCT05577663
Title: Guided Bone Regeneration in Alveolar Socket Using a Synthetic Resorbable Membrane. a Randomized Controlled Trial
Brief Title: Guided Bone Regeneration in Alveolar Socket
Acronym: GBR_socket
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Danae A. Apatzidou, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTh-79/13-02-2020
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-04

CONDITIONS: Alveolar Bone Resorption
Keywords: socket seal; randomized controlled clinical trial; alveolar ridge preservation; polylactic-glycolic acid membrane; free gingival graft; spontaneous healing
MeSH Terms: conditions — Remission, Spontaneous

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial having 3 parallel intervention arms for alveolar ridge preservation and prevention of future alveolar bone resorption due to volumetric changes of tissues post-tooth extraction.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Treatment is disclosed to the examiner after all data have been collected; investigator and care provider are different individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spontaneous healing (Other): Routine treatment of the extraction socket. Extraction of the tooth and suturing of the extraction socket with resorbable suture PGA 5/0 (polygalactic acid 5/0 sutures; PGA, medipac, Greece).
  Interventions: Other: Routine treatment of the extraction socket
- Free gingival graft (Active Comparator): Extraction of the tooth, placement of a Free Gingival Graft taken from the palate and adjusted to seal the socket opening and stabilize it by resorbable sutures PGA 5/0 (polygalactic acid 5/0 sutures; PGA, medipac, Greece).
  Interventions: Procedure: Socket seal technique by a free gingival graft
- Polylactic-Glycolic Acid membrane (Experimental): Extraction of the tooth, adjustment of the Polylactic-Glycolic Acid membrane (PLGA,Tisseos®, Biomedical Tissues, Septodont, France) over the socket opening resting by 1 mm over the alveolar crest of the extraction socket. Tissues are sutured over the barrier by resorbable sutures PGA 5/0 (polygalactic acid 5/0 sutures; PGA, medipac, Greece).
  Interventions: Procedure: Socket seal technique using a synthetic resorbable membrane

INTERVENTIONS:
Other: Routine treatment of the extraction socket — Suturing of the extraction socket with resorbable suture PGA 5/0 in order to protect the blood clot
  Arms: Spontaneous healing
Procedure: Socket seal technique by a free gingival graft — Placement of a free gingival graft in the socket opening in order to protect and stabilize the blood clot followed by suturing
  Arms: Free gingival graft
Procedure: Socket seal technique using a synthetic resorbable membrane — Placement of a synthetic barrier in the socket opening in order to protect and stabilize the blood clot followed by suturing
  Arms: Polylactic-Glycolic Acid membrane

SUMMARY:
Following tooth extraction, volumetric changes in the soft and hard tissues of the extraction site are expected to occur with considerable resorption of the alveolar bone in both the vertical and the horizontal dimensions. These changes may complicate surgical implant placement and may also compromise the outcome of the prosthetic reconstruction. Various treatment approaches have been introduced aiming to preserve the dimensions of the alveolar ridge at the extraction site and facilitate optimal implant placement.

This prospective randomized controlled trial aims to determine the efficacy of alveolar ridge preservation utilizing two different socket seal approaches compared to spontaneous healing to stabilize the blood clot within the postextraction socket. Thirty-six subjects will be randomly allocated into one of the three treatment groups. Group-A: Extraction of the tooth and suturing of the extraction socket with resorbable suture PGA 5/0. Group-B: Extraction of the tooth and placement of a Free Gingival Graft stabilized with resorbable suture PGA 5/0. Group-C: Extraction of the tooth and placement of the Polylactic-Glycolic Acid membrane stabilized with resorbable suture PGA 5/0. After the initial examination for screening, subjects will be assessed at baseline-extraction day- and after 1, 2, and 6 weeks, and 3 months. The changes of the alveolar crest will be determined in height and width, in addition to volumetric changes in the soft tissues, and the width of keratinized tissues. The wound healing process will be visually assessed.

DETAILED DESCRIPTION:
This prospective randomized controlled trial aims to determine the effectiveness of two different approaches of the "socket seal technique" for the preservation of the soft and hard tissues at the extraction site by utilizing a free gingival graft (FGG) or a PLGA membrane to stabilize the blood clot within the extraction socket compared with spontaneous healing of the tissues.

Primary outcome variable of the study will be alveolar bone changes in height buccally and palatally.

Secondary outcome variables: Alveolar bone changes in width, Mucosa thickness changes, Wound healing visual assessment, Width of keratinized tissues.

Materials and methods Thirty-six subjects will be randomly allocated into one of the three treatment groups based on computer-generated lists using a "block-design". Each patient contributes with one study site.

Study groups:

Group-A: Extraction of the tooth and suturing of the extraction socket with resorbable suture PGA 5/0.

Group-B: Extraction of the tooth, deepithelialization of the gingival colar of the socket, placement of a Free Gingival Graft taken from a standardized location of the palate adjusted to seal the socket opening and then stabilize it by resorbable suture PGA 5/0.

Group-C: Extraction of the tooth, retraction of mucoperiosteal flaps by 2 mm at the opening of the socket using a microsurgical elevator followed by adjustment of the Polylactic-Glycolic Acid membrane over the socket opening resting by 1 mm over the alveolar crest of the extraction socket. Tissues are sutured over the barrier by resorbable suture PGA 5/0.

Timeline of the study/Clinical procedures:

First visit - initial examination - (1 week before the surgery)

* Suitability of subjects
* Consent form; Randomization of the patient
* Radiographic examination (Long-cone paralleling technique using a digital sensor attached to a custom-made silicone bite block for reproducible radiographs)
* Intra-oral photography
* Impression of the examined area in order to create a reference stent to reproduce in a standard manner the clinical/radiographic measurements.
* Full mouth scaling; oral hygiene instructions

Second visit - Baseline - T0

* Clinical measurements with the use of the reference stent of:

  (i) The width of keratinized tissues with the use of a periodontal probe (Hu-Friedy XP-23/QW) (ii) The thickness of mucosa with the use of an ultrasonic device SDM (iii) The buccal osseous plate in relation to the gingival margin with a periodontal probe.
* Extraction of the tooth in a standardized way to minimize trauma; Post-surgical instructions will be given to the patient. Treatment of the extraction site accordingly to randomized treatment approach (Group-A, -B, -C).

  (i) Radiographic examination: (ii) Standardized intraoral x-ray and standardized CBCT (with the use of a reference stent)

Third visit - T1 - (1 week after the surgery)

* Evidence of healing
* Intra-oral photography

Fourth visit - T2 - (2 weeks after the surgery)

* Evidence of healing
* Removal of sutures
* Intra-oral photography

Fifth visit - T3 - Re-evaluation (6 weeks after the surgery)

* Intra-oral photography
* Width of keratinized tissues with the use of periodontal probe (Hu-Friedy XP-23/QW)
* Thickness of mucosa determined by the ultrasonic device SDM in the aforementioned standardized points with the use of the reference stent.
* Radiographic examination (The long-cone paralleling technique will be used at a distance of 10 cm between the X-ray head and the digital sensor which is attached to a custom-made silicone bite block for reproducible radiographs.)

Sixth visit - T4 - Final evaluation (3 months after the extraction)

* Intra-oral photography
* Record of periodontal plaque index (Pl) and bleeding on probing (BoP) at the adjacent teeth with the use of periodontal probe (Hu-Friedy XP-23/QW).
* Record of the width of keratinized tissues with the use of periodontal probe (Hu-Friedy XP-23/QW) and the thickness with the use of the ultrasonic device SDM in the aforementioned standardized points with the use of the reference stent.
* Radiographic examination with standardized intraoral x-ray and CBCT (with the use of the reference stent)

ELIGIBILITY:
Inclusion Criteria:

* Referrals for a single tooth extraction
* Periodontal destruction less than 50% of tooth support
* Signed inform consent form

Exclusion Criteria:

* Systematic diseases, contradicting surgical procedures and compromise wound healing (i.e. uncontrolled diabetes)
* Medication that interferes with bone metabolism
* Pregnancy or lactation
* Multiple extractions
* Absence of adjacent teeth
* Loss of buccal bone, either due to periodontal disease or because of traumatic extraction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Osseous changes in height of the alveolar ridge | Clinically: immediately after tooth extraction(baseline), 6 weeks and 3 months after the extraction. CBCT: immediately after the extraction and 3 months after the extraction
  The height of the alveolar ridge will be measured at standardized points distal, mesial and buccal/ palatal/ lingual at standardized points with the use of a reference stent by a CBCT.
Osseous changes in width of the alveolar ridge | Immediately after the extraction(baseline) and 3 months after the extraction
  The width of the alveolar ridge will be measured distal, mesial and buccal/ palatal/ lingual at standardized points with the use of a reference stent by a CBCT.

SECONDARY OUTCOMES:
Mucosa thickness changes | Baseline, 6 weeks and 3 months after the extraction
  The thickness of the keratinized tissues will be determined with the use of an ultrasonic device SDM (Austenal Medizintechnik, Koln, Germany) for recording soft tissue thickness at standardized points with the use of a reference stent.
Width of keratinized tissues | Baseline, 6 weeks and 3 months after the extraction
  The width of the keratinized tissues will be determined on the buccal aspect by a manual periodontal probe (Hu-Friedy XP-23/QW) in a standardized way by the use of a reference stent at three time-points. All recordings will be transferred to a digital caliber
Wound healing | 1 and 2 weeks after the extraction
  Visual assessment of healing

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School, Aristotle University, Dept of Preventive Dentistry, Periodontology and Implant Biology, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Overall data but not on an individual basis will be disclosed and shared

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Farmer M, Darby I. Ridge dimensional changes following single-tooth extraction in the aesthetic zone. Clin Oral Implants Res. 2014 Feb;25(2):272-7. doi: 10.1111/clr.12108. Epub 2013 Jan 25. PMID 23346895
- [Background] Maiorana C, Poli PP, Deflorian M, Testori T, Mandelli F, Nagursky H, Vinci R. Alveolar socket preservation with demineralised bovine bone mineral and a collagen matrix. J Periodontal Implant Sci. 2017 Aug;47(4):194-210. doi: 10.5051/jpis.2017.47.4.194. Epub 2017 Aug 11. PMID 28861284
- [Background] Prato GP, Cairo F, Tinti C, Cortellini P, Muzzi L, Mancini EA. Prevention of alveolar ridge deformities and reconstruction of lost anatomy: a review of surgical approaches. Int J Periodontics Restorative Dent. 2004 Oct;24(5):434-45. doi: 10.11607/prd.00.0602. PMID 15506024
- [Background] Jung RE, Siegenthaler DW, Hammerle CH. Postextraction tissue management: a soft tissue punch technique. Int J Periodontics Restorative Dent. 2004 Dec;24(6):545-53. PMID 15626317
- [Background] Annunziata M, Guida L, Nastri L, Piccirillo A, Sommese L, Napoli C. The Role of Autologous Platelet Concentrates in Alveolar Socket Preservation: A Systematic Review. Transfus Med Hemother. 2018 May;45(3):195-203. doi: 10.1159/000488061. Epub 2018 May 3. PMID 29928175